CLINICAL TRIAL: NCT05069311
Title: Effects of Multimodal Analgesia on Monocyte Chemoattractant Protein-1, Brain-derived Neurotrophic Factor, and RNA-124 Micro to Acute Pain in Patients Who Underwent Hysterectomy
Brief Title: Effects of Multimodal Analgesia on Serum MCP-1, BDNF, and MiRNA-124 in Hysterectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Christopher Ryalino, MD, Principal Investigator, Udayana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNUD-CTR-FK240921-001
Record Dates: First submitted 2021-09-23; First posted 2021-10-06 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Inflammation; Inflammatory Response; Acute Pain; Chronic Pain
MeSH Terms: conditions — Inflammation; Acute Pain; Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hysterectomy (Experimental): Patients who undergo surgical hysterectomy that fits inclusion and exclusion criteria
  Interventions: Drug: Multimodal analgesia; Drug: Conventional intravenous analgesia

INTERVENTIONS:
Drug: Multimodal analgesia — Multimodal analgesia includes the combination of:
  1. morphine given by PCA (patient-controlled analgesia) at 1 mg/dose
  2. bupivacaine 0.25% and dexmedetomidine 0.5 mcg/mL (total volume of 10 mL) by epidural-catheter bolus given preoperatively
  3. bupicavaine 0.125% and dexmedetomidine 0.5 mcg/mL at a 5 mL/hour rate per epidural-catheter given intraoperatively
  4. bupivacaine 0.1% and dexmedetomidine 0.5 mcg/mL given by programmed intermittent epidural bolus (PIEB), set to be delivered every one-hour
  5. etericoxib 90 mg per oral give two-hours before surgery and then continued until three days post-surgery
  6. paracetamol 1 g (intravenously) given on the day of the surgery, continued at 10 mg/kg dose every 8 hours until three days post-surgery
  Other Names: Group M
Drug: Conventional intravenous analgesia — Standard analgesia includes fentanyl 2 mcg/kg (bolus) and morphine given by PCA (patient-controlled analgesia) at 1 mg/dose
  Other Names: Group C

SUMMARY:
The inflammatory process is the main mechanism in the occurrence of acute postoperative pain. It is also the main risk for the development of acute pain into persistent pain. Inflammation occurs in the process of peripheral sensitization and central sensitization with various inflammatory mediators. Postoperatively, there will be proliferation and activation of microglia and astrocytes which will then activate inflammatory receptors and signaling cascades of neurotransmitters, cytokines, and chemokines. There has been a lot of clinical research evidence that multimodal analgesia can adequately treat acute pain and can prevent the development of acute postoperative pain into persistent pain and chronic postoperative pain, but the molecular mechanisms are not fully understood.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective hysterectomy
* American Society of Anesthesiologists (ASA) physical status 1 to 3

Exclusion Criteria:

* allergy to studied drugs
* history of chronic pain
* history of hepatitis, depression, peptic ulcer, or acute myocardial infarction
* receive intraoperative massive blood transfusion
* prolonged coagulation
* body mass index >35 kg/m2
* patients with neurological deficits
* taking anti-platelet medications

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Preoperative MCP-1 | 1-hour before surgery
  serum level of MCP-1
Preoperative BDNF | 1-hour before surgery
  serum level of BDNF
Preoperative MiRNA-124 | 1-hour before surgery
  serum level of MiRNA-124
Postoperative MCP-1 | 48-hours after surgery
  serum level of MCP-1
Postoperative BDNF | 48-hours after surgery
  serum level of BDNF
Postoperative MiRNA-124 | 48-hours after surgery
  serum level of MiRNA-124

CONTACTS AND LOCATIONS:
Locations (1):
- Sanglah General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided